CLINICAL TRIAL: NCT02845648
Title: The Ability to Awaken Can be Improved With Control of Lower Urinary Tract Symptoms in Children With Nonmonosymptomatic Enuresis
Brief Title: Ability to Awaken in Nonmonosymptomatic Enuresis
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kwanjin Park, professor, Seoul National University Hospital
Other Study IDs: SNUHPEDURO-01
Record Dates: First submitted 2016-07-12; First posted 2016-07-27 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Enuresis, Nocturnal, 2 (Disorder)
Keywords: anticholinergics; awakener
MeSH Terms: conditions — Enuresis | interventions — Cholinergic Antagonists; Solifenacin Succinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: anticholinergic — Initial anticholinergic therapy to all patients
  Other Names: Vesicare; BUP-4

SUMMARY:
To evaluate the effect of controlling lower urinary tract symptoms (LUTS) with anticholinergics on improving the ability to awaken (AA) in children with nonmonosymptomatic enuresis and evaluate the potential implication of improved AA for treatment response prediction.

DETAILED DESCRIPTION:
Nocturnal enuresis is associated with three main etiologies, including nocturnal polyuria secondary to abnormal anti-diuretic hormone levels, low bladder capacity related to lower urinary tract dysfunction, and sleep disorders causing problems in arousal. Among them, the association between enuresis and lower urinary tract symptoms (LUTS) has gained importance. If these two conditions coexist, the diagnosis is nonmonosymptomatic enuresis (NME). The reported prevalence of LUTS among enuretic patients ranges widely from 21% to 99%. Moreover, it was reported that spontaneous resolution can be prolonged, and some cases of NME are likely to become refractory if treated like monosymptomatic enuresis (ME) cases. A possible explanation for this may be the presence of bladder dysfunction that is not addressed properly by the standard treatment of ME. However, this explanation is only speculative.

By showing a paradoxical increase in light sleep and higher cortical arousal index in enuretic children with reduced bladder capacity, one of the reason for impaired ability to awaken (AA) in enuretic patients may lie in the chronic stimulation of the bladder. This kind of bladder dysfunction leading to an abnormal bladder-brain dialogue has been further elaborated by an experiment showing brain dysfunction in the ventrolateral periaqueductal gray matter as a result of the experimental reduction of the bladder capacity. If this is true for enuretic children, we may be able to improve arousal (improved AA) by increasing their bladder capacity.

Based on this hypothesis, the present study aimed to evaluate to the effects of anticholinergic therapy with standard urotherapy on improvement of AA and show the effect of improved AA on treatment response in children with NME.

ELIGIBILITY:
Inclusion Criteria:

* primary nonmonosymptomatic enuresis who received initial anticholinergic therapy

Exclusion Criteria:

* any urological abnormalities including neuropathic bladder

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with primary nonmonosymptomatic enuresis who received initial anticholinergic therapy
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of ability to awaken | Baseline, 3 months and 6 months
  Visual analog scale for ability to awaken (grade 1 = wake up before bed-wetting, grade 2 = wake up after bed-wetting, and grade 3 = failure of waking up around bed-wetting)

SECONDARY OUTCOMES:
Change of enuresis events | Baseline, 3 months and 6 months
  enuresis events as assessed by modified dysfunctional voiding symptoms score questionnaire (number of wet-nights per week, range 0 to 7)

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin PArk, Pf., Study Chair — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No